CLINICAL TRIAL: NCT00855621
Title: Prognostic Factors in Parkinson's Disease Patients Treated With Deep Brain Stimulation of the Subthalamic Nucleus (STN-DBS) - a Prospective Randomized Double-blind Study (The NORSTIM Study)
Brief Title: Effects of Deep Brain Stimulation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Mathias Toft, Consultant neurologist, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RRHF-PD-01
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: deep brain stimulation; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single microelectrode (Active Comparator): Surgical procedure performed using single microelectrode recording guidance intraoperatively
  Interventions: Procedure: Deep brain stimulation of the subthalamic nucleus
- Multiple microelectrode (Active Comparator): Surgical procedure performed using multiple microelectrode recording guidance intraoperatively
  Interventions: Procedure: Deep brain stimulation of the subthalamic nucleus

INTERVENTIONS:
Procedure: Deep brain stimulation of the subthalamic nucleus — Chronic bilateral deep brain stimulation in the nucleus subthalamicus is performed using the most effective of four electrode contacts identified during testing of stimulation settings. Stimulation settings will be variable and adjusted according to the symptoms of each individual patient. Stimulation parameters will be recorded at each individual examination. Dopaminergic and other necessary medication will be given according to the need of each patient.

SUMMARY:
The purpose of this study is to identify factors predicting good results in patients treated with deep brain stimulation for Parkinson's disease. The study includes a comparison of two surgical methods used to provide this therapy.

DETAILED DESCRIPTION:
The study will prospectively examine the effects of deep brain stimulation of the subthalamic nucleus (STN-DBS) on motor function, quality of life and cognitive function in Parkinson's disease (PD) patients treated at Rikshospitalet University Hospital. The aim is to identify which factors that predict good treatment outcome, in order to improve patient selection of this generally highly effective, but specialized and expensive treatment.

The study has several aims:

1. Randomized double-blind evaluation of the impact of using single vs. multiple electrode-recordings to guide electrode placement.
2. To identify factors predicting good effect on motor function and improvements of quality of life after deep brain stimulation of the subthalamic nucleus.
3. To identify cognitive and psychiatric changes related to deep brain stimulation of the subthalamic nucleus
4. To study social functioning of patients after STN-DBS and quality of life of patient caregivers

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Symptoms ≥ 5 years
* Severity of Parkinson's disease ≥ 20 points in UPDRS motor scale (scale 0-108) in OFF medication state
* Marked fluctuations of motor symptoms AND/OR troublesome dyskinesias AND/OR severe tremor AND/OR intolerable side-effects of dopaminergic drugs
* Failure of medical treatment to sufficiently control symptoms
* L-dopa responsive symptoms with ≥30% reduction in UPDRS motor score in drug ON state compared to OFF state OR severe l-dopa unresponsive tremor

Exclusion Criteria:

* Previous surgery for Parkinson's disease
* Marked axial motor symptoms unresponsive to treatment with l-dopa
* Dementia (Mattis dementia rating scale < 130).
* Patient suffering from untreated moderate or major depression or anxiety disorder
* Presence of other psychiatric disorder preventing necessary co-operation
* Brain MRI showing marked atrophy or white matter changes
* Increased risk of bleeding
* Presence of medical illness with short life expectancy
* Other surgical contra-indications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the motor score of the New-UPDRS (part III) OFF medication | 12 months

SECONDARY OUTCOMES:
Change from baseline of Clinical Dyskinesia Rating Scale score | 12 months
Change from baseline in ADL function (UPDRS part II) | 12 months
Change from baseline in Mattis Dementia Rating Scale score | 12 months
Change in social functioning (Social adjustment scale-SR) | 12 months
Change from baseline in caregivers quality of life (Scale of Caregivers Quality of Life) | 12 months
Change from baseline of self-reported health-related quality of life (PDQ-39 Summary Index) | 12 months
Frequency of new or worsened psychiatric symptoms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Espen Dietrichs, MD, PhD, Principal Investigator — Department of Neurology, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Bjerknes S, Toft M, Konglund AE, Pham U, Waage TR, Pedersen L, Skjelland M, Haraldsen I, Andersson S, Dietrichs E, Skogseid IM. Multiple Microelectrode Recordings in STN-DBS Surgery for Parkinson's Disease: A Randomized Study. Mov Disord Clin Pract. 2018 May 8;5(3):296-305. doi: 10.1002/mdc3.12621. eCollection 2018 May-Jun. PMID 30009214